CLINICAL TRIAL: NCT00250809
Title: CVC Pros and Cons of Scheduled Triple-lumen Central Venous Catheter Exchange: A Prospective Controlled Randomized Study
Brief Title: Scheduled Triple-lumen Central Venous Catheter Exchange: A Prospective Controlled Randomized Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This does not meet the requirement date to be entered into CT.gov.
Sponsor: University of New Mexico (Other)
Responsible Party: Harriet Smith, MD; Principal Investigator, University of New Mexico - CRTC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVC
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Other Female Genital; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Placement of a central venous catheter — Placement of a central venous catheter

SUMMARY:
CVC Pros and Cons of scheduled Triple-lumen Central Venous Catheter Exchange: A Prospective Controlled Randomized Study

ELIGIBILITY:
Inclusion Criteria:

1. Patients who require the placement of a central venous catheter for medical purposes and have an absence of infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1994-03 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Pros and Cons of scheduled Triple-lumen Central Venous Catheter Exchange | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Smith, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States